CLINICAL TRIAL: NCT03229278
Title: A Phase I Study to Evaluate the Safety of Trigriluzole (FC-4157/BHV-4157) in Combination With PD-1 Blocking Antibodies
Brief Title: Trigriluzole With Nivolumab and Pembrolizumab in Treating Patients With Metastatic or Unresectable Solid Malignancies or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Biren Saraiya, MD, Assistant Professor, Medical Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 051707; NCI-2017-01155 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000453; Pro20170000453 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Renal Cell Cancer; Recurrent Bladder Carcinoma; Recurrent Classical Hodgkin Lymphoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Renal Cell Carcinoma; Stage III Bladder Cancer; Stage III Lymphoma; Stage III Non-Small Cell Lung Cancer AJCC v7; Stage III Renal Cell Cancer; Stage III Skin Melanoma; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIA Skin Melanoma; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Bladder Cancer; Stage IV Lymphoma; Stage IV Non-Small Cell Lung Cancer AJCC v7; Stage IV Renal Cell Cancer; Stage IV Skin Melanoma; Stage IVA Bladder Cancer; Stage IVB Bladder Cancer; Unresectable Head and Neck Squamous Cell Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trigriluzole, nivolumab, pembrolizumab) (Experimental): Patients receive trigriluzole PO QOD, BID, QAM or QHS on days -14 to -1. Patients then receive nivolumab IV over 60 minutes every 2 weeks beginning week 1 and trigriluzole PO QOD, BID, QAM or QHS. Once the MTD of trigriluzole with nivolumab is identified, patients receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and trigriluzole PO. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzyme Inhibitor Therapy; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Enzyme Inhibitor Therapy — Given trigriluzole PO
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial studies the best dose and side effects of trigriluzole in combination with nivolumab and pembrolizumab in treating patients with solid malignancies or lymphoma that has spread to other places in the body or cannot be removed by surgery. Trigriluzole may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as nivolumab and pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving trigriluzole in combination with nivolumab and pembrolizumab may work better at treating patients with solid malignancies or lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to determine the safety of trigriluzole in combination with PD-1 inhibiting antibodies, and to define a maximum tolerated dose (MTD) of trigriluzole in combination therapy.

SECONDARY OBJECTIVES:

I. To characterize the efficacy of the combination therapy. II. To identify markers of response to trigriluzole in the tumor microenvironment.

OUTLINE: This is a dose-escalation study of trigriluzole.

Patients receive trigriluzole orally (PO) every other day (QOD), twice daily (BID), every morning (QAM) or every bedtime (QHS) on days -14 to -1. Patients then receive nivolumab intravenously (IV) over 60 minutes every 2 weeks beginning week 1 and trigriluzole PO QOD, BID, QAM or QHS. Once the MTD of trigriluzole with nivolumab is identified, patients receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and trigriluzole PO. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid malignancy or lymphoma that is metastatic or unresectable
* There is reasonable expectation of response to pembrolizumab or nivolumab, and one of the drugs is available from the commercial supply; this includes (but is not limited to) the following tumor types: melanoma, non-small cell lung cancer, renal cell carcinoma, squamous cell carcinoma of the head and neck, bladder cancer, and classic Hodgkin lymphoma
* The patient must have failed at least one line of standard treatment, with the following exceptions in which a PD-1 antibody is Food and Drug Administration (FDA) approved in the first-line setting:

  * Melanoma patients
  * Non-small cell lung cancer patients without EGFR or ALK genomic tumor aberrations whose tumors have high PD-L1 expression (tumor proportion score [TPS] >= 50%) as determined by an FDA-approved test
* Patients must give informed consent
* Prior chemotherapy, immunotherapy, radiotherapy or major surgery (including radiation therapy or surgery for treatment of brain metastases) must be completed at least 3 weeks before study entry; prior PD-1 or PD-L1 therapy is acceptable
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin > 8.0 mg/dL (without transfusion in the preceding 7 days)
* Platelets >= 70,000 /uL
* Total bilirubin within normal institutional limits (patients with Gilbert's syndrome must have a total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 2 X institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 X institutional ULN
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm by computed tomography (CT) scan, positron emission tomography (PET)/CT scan, magnetic resonance imaging (MRI) or caliper/ruler measurement by clinical exam; lymph nodes: to be considered pathologically enlarged and measurable, a lymph node must be >= 15 mm in short axis when assessed by CT scan; lesions that have been radiated in the advanced setting cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy
* Ability to swallow pills

Exclusion Criteria:

* Systemic immunosuppressive medications such as steroids; the following steroid formulations are permitted: intranasal, intra-articular, and inhaled steroids
* History of immune-related adverse event from prior immunotherapy treatment that has not improved to grade 0-1; subjects with grade 2 hypothyroidism and grade 2 adrenal insufficiency requiring continued medical treatment may enroll provided that they are asymptomatic and stable on their dose of hormone replacement
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient?s ability to complete the study, at the discretion of the investigator, including active autoimmune disease requiring treatment within the past 30 days
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption)' physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Second primary malignancy, except those second primary malignancies that are not considered to be competing causes of death in the opinion of the treating investigator; examples include: in situ carcinoma of the cervix, adequately treated non-melanoma carcinoma of the skin, or other malignancy treated at least 5 years previously with no evidence of recurrence
* Patients with active, untreated central nervous system (CNS) metastases will be excluded from this clinical trial; patients who have brain metastases that been treated with radiation therapy or surgery will be required to have a washout period of at least 3 weeks prior to study entry, must be neurologically asymptomatic, and must not require systemic steroids
* Women of child-bearing potential and men must agree to use adequate contraception prior to the start of treatment, for the duration of treatment, and for 5 months after last dose of study treatment
* Patients with immune deficiency have impaired immune responses, therefore, known human immunodeficiency virus (HIV)-positive patients are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biren Saraiya, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179
- [Derived] Silk AW, Saraiya B, Groisberg R, Chan N, Spencer K, Girda E, Shih W, Palmeri M, Saunders T, Berman RM, Coric V, Chen S, Zloza A, Vieth J, Mehnert JM, Malhotra J. A phase Ib dose-escalation study of troriluzole (BHV-4157), an oral glutamatergic signaling modulator, in combination with nivolumab in patients with advanced solid tumors. Eur J Med Res. 2022 Jul 2;27(1):107. doi: 10.1186/s40001-022-00732-w. PMID 35780243

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO): Cohort 1: Participants were administered 240 mg of Nivolumab every two weeks, via intravenous catheter (IV), for 2 weeks, and Trigriluzole 140 mg (PO), with one year of follow-up after the start of treatment.
  Once the MTD of Trigriluzole with nivolumab is identified, participants receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and Trigriluzole PO. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
- Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID): Cohort 2: Participants were administered 240 mg of Nivolumab every two weeks, via intravenous catheter (IV), for 2 weeks, and Trigriluzole 140 mg (PO) Twice a day (BID), with one year of follow-up after the start of treatment.
  Once the MTD of Trigriluzole with nivolumab is identified, participants receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and Trigriluzole PO. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
- Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg: Cohort 3: Participants were administered 240 mg of Nivolumab every two weeks, via intravenous catheter (IV) and Trigriluzole 140 mg (PO) once a day in the morning (QAM) and 280mg PO every night at bedtime (QHS), with one year of follow-up after the start of treatment.
  Once the MTD of Trigriluzole with nivolumab is identified, participants receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and Trigriluzole PO. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
- Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID: Cohort 4: Participants were administered 240 mg of Nivolumab every two weeks, via intravenous catheter (IV) and Trigriluzole 140 mg (PO) once a day in the morning (QAM) and 280mg PO every night at bedtime (QHS), with one year of follow-up after the start of treatment.
  Once the MTD of Trigriluzole with nivolumab is identified, participants receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and Trigriluzole 200mg PO BID. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Started | 3 | 6 | 3 | 2
Completed | 3 | 6 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID | Total
Number analyzed (Participants) | 3 | 6 | 3 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 0 | 5
  >=65 years | 2 | 3 | 2 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 0 | 6
  Male | 2 | 2 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 3 | 6 | 2 | 1 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD))/Recommended Phase 2 Dose of Trigriluzole
Description: The MTD of trigriluzole in combination with nivolumab will be identified. The MTD will then be tested in combination with pembrolizumab using the same escalate/de-escalate/stay rules. Data on the adverse event type, severity and frequency will be recorded.
Time Frame: Four weeks
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least 1 dose of Trigriluzole (140 mg or 280mg ) in combination with Nivolumab (240mg IV)
Arm/Group | All Participants
Number analyzed (Participants) | 14
mg | 420

2. Secondary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLT)
Description: A DLT was any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE 3.0) that was possibly Trigriluzole or Nivolumab related. CTCAE 3.0 Grade 3 is a severe AE and Grade 4 is a life- threatening or disabling AE. DLTs were collected to determine the Maximum-Tolerated Dose (MTD), which is defined as the dose level below the dose at which 33% of participants experienced a DLT.
Time Frame: Four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 3 | 6 | 3 | 2
Participants | 0 | 0 | 1 | 2

3. Secondary Outcome: Objective Response Rate Assessed According to Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Continuous variables will be presented by summary statistics (such as mean, median, standard error and 95% confidence intervals [CI]) and the categorical variables by frequency distributions (i.e., frequency counts, percentages and 95% CI).
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID: Cohort 4: Participants were administered 240 mg of Nivolumab every two weeks, via intravenous catheter (IV) and Trigriluzole 140 mg (PO) once a day in the morning (QAM) and 280mg PO every night at bedtime (QHS), with one year of follow-up after the start of treatment.
  Once the MTD of Trigriluzole with nivolumab is identified, participants receive pembrolizumab IV over 30 minutes every 3 weeks beginning week 1 and Trigriluzole 200mg PO BID. Treatment repeats for up to 1 year in the absence of disease progression or unacceptable toxicity.
Arm/Group | Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 14
percentage of participants | 7 [0.2 to 33.9]

4. Secondary Outcome: Overall Survival
Description: Continuous variables will be presented by summary statistics (such as mean, median, standard error and 90% CI) and the categorical variables by frequency distributions (i.e., frequency counts, percentages and 90% CI).
Time Frame: Up to 3 years
Population: no data collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Next Therapy or Death
Description: as for outcome 4
Time Frame: Up to 3 years
Population: No data collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Freedom From New Metastases
Description: as for outcome 4
Time Frame: Up to 3 years
Population: No Data collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Landmark Survival Rates at 1 Year
Description: as for outcome 4
Time Frame: 1 year
Population: data not collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Landmark Survival Rate at 2 Years
Description: as for outcome 4
Time Frame: 2 years
Population: No data collected.
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Duration of Response for Responding Patients
Description: as for outcome 4
Time Frame: Up to 3 years
Population: data not collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Progression Free Survival
Description: as for outcome 4
Time Frame: Up to 3 years
Population: Data not collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Time to Treatment Failure
Description: as for outcome 4
Time Frame: Up to 3 years
Population: Data not collected
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline and up to three years after the last dose
Description: A DLT was any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE 3.0) that was possibly Trigriluzole or Nivolumab related. CTCAE 3.0 Grade 3 is a severe AE and Grade 4 is a life- threatening or disabling AE. DLTs were collected to determine the Maximum-Tolerated Dose (MTD), which is defined as the dose level below the dose at which 33% of participants experienced a DLT.
Arm/Group | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/6 | 2/3 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/6 | 0/3 | 2/14
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) (N=3) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) (N=6) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg (N=3) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID (N=14)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg Taken by Mouth Daily (PO) (N=3) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg PO Twice a Day (BID) (N=6) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 140 mg /280mg (N=3) | Experimental: Nivolumab 240mg IV Every 2 Weeks - Trigriluzole 280mg PO BID (N=14)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (14) | 2 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (7) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Gastrointestinal disorders - (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (12)
Pain (General disorders) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (3) | 1 (1) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (2) | 1 (1) | 2 (4)
Lipase increased (Investigations) | 1 (1) | 4 (7) | 1 (1) | 1 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (3) | 2 (3) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Platelet count decreased (Investigations) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 1 (1) | 2 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 2 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 2 (3) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03229278/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03229278/ICF_000.pdf